CLINICAL TRIAL: NCT04790201
Title: Adaptation of the Friendship Bench Counseling Intervention to Improve Mental Health and HIV Care Engagement Outcomes Among People Living With HIV Who Inject Drugs in Vietnam
Brief Title: Friendship Bench Adaptation to Improve Mental Health & HIV Care Engagement Outcomes Among PLWH and PWID in Vietnam
Acronym: VITAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Hanoi Medical University (Other); The Friendship Bench Trust (Other); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20-1689; R34DA051933 (NIH); IGHID 12028 (Other: UNC-CH)
Record Dates: First submitted 2021-02-18; First posted 2021-03-10 (Actual); Results first posted 2024-08-13 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-05

CONDITIONS: HIV Infections; Behavioral Symptoms; Depression; Anxiety; Opioid-use Disorder; Virus Infection; Immune System Diseases; Opioid Dependence
MeSH Terms: conditions — HIV Infections; Behavioral Symptoms; Depression; Anxiety Disorders; Opioid-Related Disorders; Virus Diseases; Immune System Diseases

STUDY DESIGN:
Intervention Model Description: Three-arm individually randomized trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Friendship Bench Delivered by Professional Counselor (Experimental): Participants seeking HIV and/or MMT services at participating clinics in Hanoi, Vietnam will be enrolled in this study arm during study recruitment. Individuals enrolled in this arm will initiate FB with a professional counselor. Individuals enrolled in this arm will receive 6 weekly counseling sessions per the adapted FB protocol (Aim 1).
  Interventions: Behavioral: Friendship Bench Delivered by Professional Counselor
- Friendship Bench Delivered by Lay Counselor (Experimental): Participants seeking HIV and/or MMT services at participating clinics in Hanoi, Vietnam will be enrolled in this study arm during study recruitment. Individuals enrolled in this arm will initiate FB with a trained lay counselor. Individuals enrolled in this arm arm will receive 6 weekly counselling sessions per the adapted FB protocol (Aim 1).
  Interventions: Behavioral: Friendship Bench Delivered by Lay Counselor
- Enhanced Usual Care (Active Comparator): Participants seeking HIV and/or MMT services at participating clinics in Hanoi, Vietnam will be enrolled in this study arm during study recruitment. Enhanced usual care will include general training of the HIV providers and clinics about CMD identification and management, and feedback to the HIV provider of the status of their enrolled patient to allow follow-up per the clinic's standard care.
  Interventions: Behavioral: Enhanced Usual Care

INTERVENTIONS:
Behavioral: Friendship Bench Delivered by Professional Counselor — Participants randomized to this arm will receive the Friendship Bench protocol delivered by a professional counselor.
  Arms: Friendship Bench Delivered by Professional Counselor
Behavioral: Friendship Bench Delivered by Lay Counselor — Participants randomized to this arm will receive the Friendship Bench protocol delivered by a trained lay counselor.
  Arms: Friendship Bench Delivered by Lay Counselor
Behavioral: Enhanced Usual Care — Enhanced usual care (EUC) will include general training of the HIV providers and clinics about CMD identification and management, and feedback to the HIV provider of the status of their enrolled patient to allow follow-up per the clinic's standard care. Information will be collected in follow-up interviews to characterize the care that patients receive. These activities will occur in all three arms, but they are the only activities in the EUC arm.
  Arms: Enhanced Usual Care

SUMMARY:
This project will adapt and pilot a feasible and effective problem-solving therapy designed for low-resource settings to address common mental disorders like depression and anxiety - the Friendship Bench- in a Vietnamese population of individuals living with HIV who also have opiate use disorder. The Friendship Bench approach has the potential to make an important contribution to address CMDs and reduce barriers to HIV treatment success among people living with HIV (PLWH) with Opioid Use Disorder (OUD), a critical population driving the HIV epidemic in Vietnam and many Southeast Asian countries. This proposal will generate critical evidence for designing a fully powered clinical trial to test the investigation team's adapted FB protocol in improving HIV, mental health, and drug use treatment outcomes for this vulnerable population.

DETAILED DESCRIPTION:
Injection drug use is the primary driver of the HIV epidemic in Southeast Asia. In 2017, the HIV prevalence among people who inject drugs (PWID) in Southeast Asia was 15%. PWID, most of whom have OUD, who are living with HIV have low rates of retention in care, antiretroviral therapy (ART) initiation, and viral suppression. PWID also experience high rates of HIV-related and all-cause mortality. Common mental disorders (CMDs), including depressive, anxiety, and stress-related illnesses, occur in 40-50% of PLWH and OUD. Despite serious consequences of mental illness on health and HIV progression, mental illness remains under-diagnosed and under-treated in HIV populations, especially in low- and middle-income countries (LMICs), such as many countries in Southeast Asia.

To respond to the great need for mental health treatment in low- and middle-income countries, the global mental health field has focused on developing task-shifting and integration approaches that equip non-specialists to deliver evidence-based mental health interventions at scale. However, such task shifting interventions to address CMDs have received limited attention in Southeast Asia among OUD. Vietnam, with its high prevalence of PLWH and OUD, its integration of methadone maintenance therapy (MMT) with HIV care, and its priority for developing CMD care for this population, is an ideal setting to evaluate task-shifting mental health approaches to address CMDs and improve HIV care outcomes.

The Friendship Bench (FB) is a feasible and effective task-shifting mental health intervention designed for low-resource settings that is a strong candidate to address CMDs in this population. FB is a problem solving therapy-based intervention with demonstrated effectiveness in treating CMDs among primary care patients when delivered by lay counselors. Lay counselors may effectively deliver FB to PLWH with OUD, but CMD may prove more difficult to treat in patients with OUD and require professionally trained counselors to be effective.

The investigators' objective is to complete a pilot randomized trial of 75 patients from 4 MMT clinics in Hanoi. The investigators' specific aims are: 1) To adapt the Friendship Bench (FB) protocol to be optimized for PLWH and OUD in Vietnam; and 2) To evaluate the feasibility, fidelity, and acceptability of the adapted FB as well as preliminary indicators of its impact in improving CMDs and HIV care and drug use treatment outcomes. The Friendship Bench approach has the potential to make an important contribution to address CMDs and reduce barriers to HIV treatment success among PLWH with OUD, a critical population driving the HIV epidemic in Vietnam and many Southeast Asian countries. This proposal will generate critical evidence for designing a fully powered clinical trial to test the adapted FB protocol in improving HIV, mental health, and drug use treatment outcomes for this vulnerable population.

ELIGIBILITY:
Inclusion Criteria:

Eligible individuals will meet the following criteria:

* Adult patients (18 years and older) being treated at the Methadone Maintenance Treatment (MMT) clinic
* Medical record indicates infection with HIV
* Have been screened with the Depression Anxiety Stress Scale-21 (DASS-21) which has been translated, standardized and validated in the Vietnamese population with a positive result indicating a CMD. The investigators will consider as eligible all patients with a depression subscale score ≥ 7, an anxiety subscale score ≥ 6, and/or a stress subscale score ≥ 10. Elevated depressive symptoms be present for ≥2 weeks and elevated anxiety or post-traumatic stress-related symptoms be present for ≥1 month. The investigators will consider a positive screen for any of the three categories as indicating a CMD.

Exclusion Criteria:

• Those with evidence of psychosis or bipolar disorder per the Mini International Neuropsychiatric Interview (MINI) will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2022-02-28 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bradley Gaynes, MD, MPH, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- CDC Hanoi, Hanoi, Hanoi City, Vietnam

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with the University of North Carolina at Chapel Hill (UNC).
Time Frame: 9 to 36 months following publication
Access Criteria: The investigator who proposes to use the data has approval from an IRB, IEC, or REB, as applicable, and an executed data use/sharing agreement with UNC.

REFERENCES:
- [Background] Henry JD, Crawford JR. The short-form version of the Depression Anxiety Stress Scales (DASS-21): construct validity and normative data in a large non-clinical sample. Br J Clin Psychol. 2005 Jun;44(Pt 2):227-39. doi: 10.1348/014466505X29657. PMID 16004657
- [Background] Le MTH, Tran TD, Holton S, Nguyen HT, Wolfe R, Fisher J. Reliability, convergent validity and factor structure of the DASS-21 in a sample of Vietnamese adolescents. PLoS One. 2017 Jul 19;12(7):e0180557. doi: 10.1371/journal.pone.0180557. eCollection 2017. PMID 28723909
- [Background] Tran TD, Tran T, Fisher J. Validation of the depression anxiety stress scales (DASS) 21 as a screening instrument for depression and anxiety in a rural community-based cohort of northern Vietnamese women. BMC Psychiatry. 2013 Jan 12;13:24. doi: 10.1186/1471-244X-13-24. PMID 23311374
- [Background] Mathers BM, Degenhardt L, Phillips B, Wiessing L, Hickman M, Strathdee SA, Wodak A, Panda S, Tyndall M, Toufik A, Mattick RP; 2007 Reference Group to the UN on HIV and Injecting Drug Use. Global epidemiology of injecting drug use and HIV among people who inject drugs: a systematic review. Lancet. 2008 Nov 15;372(9651):1733-45. doi: 10.1016/S0140-6736(08)61311-2. Epub 2008 Sep 23. PMID 18817968
- [Background] Degenhardt L, Peacock A, Colledge S, Leung J, Grebely J, Vickerman P, Stone J, Cunningham EB, Trickey A, Dumchev K, Lynskey M, Griffiths P, Mattick RP, Hickman M, Larney S. Global prevalence of injecting drug use and sociodemographic characteristics and prevalence of HIV, HBV, and HCV in people who inject drugs: a multistage systematic review. Lancet Glob Health. 2017 Dec;5(12):e1192-e1207. doi: 10.1016/S2214-109X(17)30375-3. Epub 2017 Oct 23. PMID 29074409
- [Background] Chesney MA. Factors affecting adherence to antiretroviral therapy. Clin Infect Dis. 2000 Jun;30 Suppl 2:S171-6. doi: 10.1086/313849. PMID 10860902
- [Background] Malta M, Strathdee SA, Magnanini MM, Bastos FI. Adherence to antiretroviral therapy for human immunodeficiency virus/acquired immune deficiency syndrome among drug users: a systematic review. Addiction. 2008 Aug;103(8):1242-57. doi: 10.1111/j.1360-0443.2008.02269.x. PMID 18855813
- [Background] Sherer R. Adherence and antiretroviral therapy in injection drug users. JAMA. 1998 Aug 12;280(6):567-8. doi: 10.1001/jama.280.6.567. No abstract available. PMID 9707152
- [Background] Jordan MR, Obeng-Aduasare Y, Sheehan H, Hong SY, Terrin N, Duong DV, Trung NV, Wanke C, Kinh NV, Tang AM. Correlates of non-adherence to antiretroviral therapy in a cohort of HIV-positive drug users receiving antiretroviral therapy in Hanoi, Vietnam. Int J STD AIDS. 2014 Aug;25(9):662-668. doi: 10.1177/0956462413516301. Epub 2013 Dec 18. PMID 24352130
- [Background] Mathers BM, Degenhardt L, Bucello C, Lemon J, Wiessing L, Hickman M. Mortality among people who inject drugs: a systematic review and meta-analysis. Bull World Health Organ. 2013 Feb 1;91(2):102-23. doi: 10.2471/BLT.12.108282. PMID 23554523
- [Background] Weber R, Huber M, Battegay M, Stahelin C, Castro Batanjer E, Calmy A, Bregenzer A, Bernasconi E, Schoeni-Affolter F, Ledergerber B; Swiss HIV Cohort Study. Influence of noninjecting and injecting drug use on mortality, retention in the cohort, and antiretroviral therapy, in participants in the Swiss HIV Cohort Study. HIV Med. 2015 Mar;16(3):137-51. doi: 10.1111/hiv.12184. Epub 2014 Aug 15. PMID 25124393
- [Background] Lappalainen L, Hayashi K, Dong H, Milloy MJ, Kerr T, Wood E. Ongoing impact of HIV infection on mortality among people who inject drugs despite free antiretroviral therapy. Addiction. 2015 Jan;110(1):111-9. doi: 10.1111/add.12736. Epub 2014 Oct 16. PMID 25203392
- [Background] Adams C, Zacharia S, Masters L, Coffey C, Catalan P. Mental health problems in people living with HIV: changes in the last two decades: the London experience 1990-2014. AIDS Care. 2016;28 Suppl 1(sup1):56-9. doi: 10.1080/09540121.2016.1146211. Epub 2016 Feb 17. PMID 26888472
- [Background] Gaynes BN, Pence BW, Eron JJ Jr, Miller WC. Prevalence and comorbidity of psychiatric diagnoses based on reference standard in an HIV+ patient population. Psychosom Med. 2008 May;70(4):505-11. doi: 10.1097/PSY.0b013e31816aa0cc. Epub 2008 Mar 31. PMID 18378865
- [Background] Bouhnik AD, Preau M, Vincent E, Carrieri MP, Gallais H, Lepeu G, Gastaut JA, Moatti JP, Spire B; MANIF 2000 Study Group. Depression and clinical progression in HIV-infected drug users treated with highly active antiretroviral therapy. Antivir Ther. 2005;10(1):53-61. PMID 15751763
- [Background] Jones DL, Waldrop-Valverde D, Gonzalez P, Mack A, Kumar AM, Ownby R, Weiss SM, Kumar M. Mental health in HIV seronegative and seropositive IDUs in South Florida. AIDS Care. 2010 Feb;22(2):152-8. doi: 10.1080/09540120903039851. PMID 19662550
- [Background] Springer SA, Chen S, Altice F. Depression and symptomatic response among HIV-infected drug users enrolled in a randomized controlled trial of directly administered antiretroviral therapy. AIDS Care. 2009 Aug;21(8):976-83. doi: 10.1080/09540120802657555. PMID 20024753
- [Background] WHO Secretariat. HIV/AIDS and mental health. World Health Institution; 2008.
- [Derived] Nong HTT, Nguyen HN, Tran HV, Cao ATV, Tran TTT, Filipowicz TR, Landrum KR, Giang LM, Verhey R, Pence BW, Gaynes BN. Providers' Experiences in Implementation of Friendship Bench: A Problem-Solving Therapy-Based Mental Health Intervention Adapted for People on Methadone Maintenance Treatment Who Live with HIV in Vietnam. AIDS Behav. 2026 Feb 6. doi: 10.1007/s10461-026-05054-0. Online ahead of print. PMID 41649734
- [Derived] Gaynes BN, Tran HV, Nong HTT, Filipowicz TR, Landrum KR, Tran TTT, Nguyen VQ, Verhey R, Nguyen HN, Giang LM, Pence BW. An Adapted Friendship Bench Counseling Intervention (FB) to Improve Mental Health and HIV Care Engagement Outcomes Among People Living with HIV (PWH) Who Inject Drugs in Hanoi, Vietnam: Results from the VITAL Pilot Randomized Controlled Trial. AIDS Behav. 2025 Jun;29(6):1761-1774. doi: 10.1007/s10461-025-04645-7. Epub 2025 Feb 2. PMID 39894853
- [Derived] Tran HV, Filipowicz TR, Landrum KR, Nong HTT, Tran TTT, Pence BW, Go VF, Le GM, Nguyen MX, Verhey R, Chibanda D, Ho HT, Gaynes BN. Stigma experienced by people living with HIV who are on methadone maintenance treatment and have symptoms of common mental disorders in Hanoi, Vietnam: a qualitative study. AIDS Res Ther. 2022 Dec 14;19(1):63. doi: 10.1186/s12981-022-00491-y. PMID 36517849
- [Derived] Tran HV, Nong HTT, Tran TTT, Filipowicz TR, Landrum KR, Pence BW, Le GM, Nguyen MX, Chibanda D, Verhey R, Go VF, Ho HT, Gaynes BN. Adaptation of a Problem-solving Program (Friendship Bench) to Treat Common Mental Disorders Among People Living With HIV and AIDS and on Methadone Maintenance Treatment in Vietnam: Formative Study. JMIR Form Res. 2022 Jul 8;6(7):e37211. doi: 10.2196/37211. PMID 35802402

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study recruitment began in February 2022. Recruitment occurred in Methadone Maintenance Treatment (MMT) clinics located in Hanoi, Vietnam.
Pre-assignment Details: Two of the randomized participants (1 in Friendship Bench delivered by Professional Counselor arm and 1 in Usual Care arm) were found to be ineligible for the study shortly after enrollment and were excluded from all analyses.
Groups:
- Enhanced Usual Care: Participants seeking HIV and/or MMT services at participating clinics in Hanoi, Vietnam will be enrolled in this study arm during study recruitment. Enhanced usual care will include general training of the HIV providers and clinics about common mental disorder (CMD) identification and management, and feedback to the HIV provider of the status of their enrolled patient to allow follow-up per the clinic's standard care.
  Enhanced Usual Care: Enhanced usual care (EUC) will include general training of the HIV providers and clinics about CMD identification and management, and feedback to the HIV provider of the status of their enrolled patient to allow follow-up per the clinic's standard care. Information will be collected in follow-up interviews to characterize the care that patients receive. These activities will occur in all three arms, but they are the only activities in the EUC arm.
Period: Overall Study
Arm/Group | Friendship Bench Delivered by Professional Counselor | Friendship Bench Delivered by Lay Counselor | Enhanced Usual Care
Started | 26 | 25 | 26
Completed | 25 | 24 | 23
Not Completed | 1 | 1 | 3
Not completed — Lost to Follow-up | 0 | 0 | 2
Not completed — Death | 0 | 1 | 0
Not completed — Protocol Violation | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Two of the randomized participants (1-Friendship Bench Delivered by Professional Counselor and 1-Enhanced Usual Care) were found to be ineligible for the study shortly after enrollment and were excluded from all analyses.
Groups:
- Total: Total of all reporting groups
Arm/Group | Friendship Bench Delivered by Professional Counselor | Friendship Bench Delivered by Lay Counselor | Enhanced Usual Care | Total
Number analyzed (Participants) | 25 | 25 | 25 | 75
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.1 (5.0) | 44.9 (7.2) | 44.9 (5.2) | 44.6 (5.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1 | 2
  Male | 25 | 24 | 24 | 73
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Vietnam | 25 | 25 | 25 | 75

OUTCOME MEASURES:

1. Primary Outcome: Total Number of Participants Who Were Eligible and Enrolled (Intervention Feasibility)
Description: This measure of feasibility will be measured as the ability to successfully enroll people living with HIV (PLWH) and opioid use disorder (OUD) with CMDs in the pilot intervention. Feasibility will be evaluated by measuring the recruitment rate (number of patients approached in order to accrue the final sample).
Time Frame: Baseline
Population: The analysis population includes the total number of people approached for study eligibility and screening. Two of the randomized participants (1-Friendship Bench Delivered by Professional Counselor and 1-Enhanced Usual Care) were found to be ineligible for the study shortly after enrollment and were excluded from all analyses.
Measure: Count of Participants; unit: Participants
Groups:
- Study Population: The study population includes the total number of study participants enrolled (regardless of assigned study arm).
Arm/Group | Study Population
Number analyzed (Participants) | 287
Participants | 75

2. Primary Outcome: Study Retention (Study Feasibility)
Description: This measure of feasibility will be measured as the ability to retain PLWH and OUD with CMDs in the pilot trial. Feasibility will be evaluated by measuring the number of participants retained in the study (number of patients enrolled at baseline who are still enrolled in the trial), through study completion.
Time Frame: Through study completion, an average of 12 months
Population: The analysis population includes the total number of eligible study participants (n=75) enrolled. Two of the randomized participants (1-Friendship Bench Delivered by Professional Counselor and 1-Enhanced Usual Care) were found to be ineligible for the study shortly after enrollment and were excluded from all analyses.
Measure: Count of Participants; unit: Participants
Arm/Group | Friendship Bench Delivered by Professional Counselor | Friendship Bench Delivered by Lay Counselor | Enhanced Usual Care
Number analyzed (Participants) | 25 | 25 | 25
Participants | 25 | 25 | 23

3. Primary Outcome: Percent of FB Sessions Attended (Intervention Feasibility)
Description: The percent of FB sessions attended by participants out of total FB sessions offered, during the target intervention duration of 6 weeks.
Time Frame: 6 weeks
Population: The analysis population includes the total number of planned intervention sessions across the two arms (FB delivered by professional counselor and FB delivered by lay counselor). Each arm had 25 participants with 6 planned, weekly sessions per participant for a total of (25*6)150 sessions per arm. The enhanced usual care arm (n=25) did not receive an intervention and are not included in the analysis population.
Measure: Number; unit: percent of FB Sessions Attended
Units Other Than Participants: Intervention Sessions
Arm/Group | Friendship Bench Delivered by Professional Counselor | Friendship Bench Delivered by Lay Counselor | Enhanced Usual Care
Number analyzed (Participants) | 25 | 25 | 0
Number analyzed (Intervention Sessions) | 150 | 150 | 0
percent of FB Sessions Attended | 100 | 100 |

4. Primary Outcome: Number of Participants Satisfied With Friendship Bench (Intervention Acceptability)
Description: The number of patients who were either very satisfied or somewhat satisfied with the FB among all participants who received the FB. Satisfaction will be measured using a single question with a 4-point Likert scale-- 1 indicates high satisfaction and 4 indicates high dissatisfaction.
Time Frame: 6 weeks
Population: The analysis population includes all participants who received the intervention [FB delivered by professional counselor (n=25) and FB delivered by lay counselor(n=25)] for a total of 50 analyzed participants. Participants who received enhanced usual care (n=25) are not included in the analysis population as they did not receive the intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Friendship Bench Delivered by Professional Counselor | Friendship Bench Delivered by Lay Counselor | Enhanced Usual Care
Number analyzed (Participants) | 25 | 25 | 0
Participants | 25 | 25 |

5. Primary Outcome: Number of Counseling Sessions Meeting Fidelity Threshold (Intervention Fidelity)
Description: The total number of FB sessions meeting or exceeding for at least 75% of the total number of fidelity checklist items assessed per session.
Time Frame: 6 weeks
Population: The analysis population includes the total number of intervention sessions across the two arms (FB delivered by professional counselor and FB delivered by lay counselor) assessed for fidelity. Each FB counselor had >=3 randomly-chosen sessions reviewed for fidelity. The FB delivered by professional counselors had n=92 sessions and the FB delivered by lay counselors has n=95 sessions. The enhanced usual care arm did not receive an intervention and are not included in the analysis population.
Measure: Number; unit: Number of sessions meeting fidelity
Units Other Than Participants: Intervention Sessions
Arm/Group | Friendship Bench Delivered by Professional Counselor | Friendship Bench Delivered by Lay Counselor | Enhanced Usual Care
Number analyzed (Participants) | 25 | 25 | 0
Number analyzed (Intervention Sessions) | 92 | 95 | 0
Number of sessions meeting fidelity | 66 | 42 |

6. Secondary Outcome: Number of Participants Achieving HIV Viral Suppression
Description: HIV viral load will be measured from clinical records, or measured and ordered by the study if no viral load is collected in the appropriate window. Viral suppression is defined as <20 copies of HIV-1 RNA per milliliter.
Time Frame: 6 months after enrollment
Population: The analysis population includes all study participants (across all 3 arms) who attended the 6-month follow-up visit and provided a sample for viral load testing. Note not all participants were able to provide a blood sample for viral load testing. The professional counselor FB arm had n=25 participants, the lay counselor FB arm had n= 24 participants, and the enhanced usual care arm had (n=23) participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Friendship Bench Delivered by Professional Counselor | Friendship Bench Delivered by Lay Counselor | Enhanced Usual Care
Number analyzed (Participants) | 25 | 24 | 23
Participants | 19 | 21 | 21

7. Secondary Outcome: Proportion of Scheduled HIV Visits That Were Attended in the 12-Month Follow-Up Period
Description: The proportion of scheduled visits in the 12-month follow-up period that are attended vs. no-shows (the "kept visit proportion"), with no-show defined as no appointment kept in the 30 days following a scheduled appointment. HIV appointment data will be abstracted from clinic records at the end of the study period.
Time Frame: Study baseline through 12 months of follow-up
Population: This analysis population includes the total number of scheduled HIV visits. The n = 25 participants in the Friendship Bench (FB) delivered by professional counselor arm contributed n= 201 HIV visits. The n = 25 participants in the FB delivered by lay counselor arm contributed n = 170 HIV appointments. The n=25 participants in the enhanced usual care arm contributed n = 179 HIV visits. The number of visits represents the total possible number of visits (regardless of attendance) in each arm.
Measure: Number; unit: proportion of scheduled visits attended
Units Other Than Participants: scheduled HIV visits
Arm/Group | Friendship Bench Delivered by Professional Counselor | Friendship Bench Delivered by Lay Counselor | Enhanced Usual Care
Number analyzed (Participants) | 25 | 25 | 25
Number analyzed (scheduled HIV visits) | 201 | 170 | 179
proportion of scheduled visits attended | 0.95 | 0.94 | 0.92

8. Secondary Outcome: Total CMD Symptoms Score for Participants
Description: CMD symptoms will be evaluated via the 21-item Depression, Anxiety, and Stress Scale (DASS-21), which consists of three subscales. Responses are ranked from 0 (Does not apply to me at all) to 3 (Applied to me very much or most of the time). All subscales are multiplied by 2. The total scale is calculated by summing the subscales, range 0-126, for depression (threshold ≥14), anxiety (threshold ≥10), and stress (threshold ≥19); higher scores indicate higher severity of symptoms.
Time Frame: 6 weeks after enrollment
Population: The analysis population includes all study participants (across all 3 arms) who attended the 6-week follow-up visit. The two intervention arms (FB by professional and lay counselors) each had n=25 participants complete the 6-week follow-up visit. The enhanced usual care arm had n=24 participants complete the 6-week follow-up visit.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Friendship Bench Delivered by Professional Counselor | Friendship Bench Delivered by Lay Counselor | Enhanced Usual Care
Number analyzed (Participants) | 25 | 25 | 24
score on a scale | 27.28 (26.4) | 23.9 (21.4) | 32.3 (22.7)

9. Secondary Outcome: Change in CMD Symptoms
Description: The change in CMD symptoms from baseline to 6 weeks in the DASS-21 total score is calculated as Baseline DASS-21 total score minus the Week 6 DASS-21 total score. CMD symptoms will be evaluated via the 21-item Depression, Anxiety, and Stress Scale (DASS-21), which consists of three subscales. Responses are ranked from 0 (Does not apply to me at all) to 3 (Applied to me very much or most of the time). All subscales are multiplied by 2. The total scale is calculated by summing the subscales, range 0-126, for depression (threshold ≥14), anxiety (threshold ≥10), and stress (threshold ≥19); higher scores indicate higher severity of symptoms.
Time Frame: Baseline, 6 weeks after enrollment
Population: The analysis population includes all study participants (across all 3 arms) who completed the 6 week followup visit. The professional counselor FB arm had n=25 participants, the lay counselor FB arm had n= 25 participants, and the enhanced usual care arm had n=24 participants.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Friendship Bench Delivered by Professional Counselor | Friendship Bench Delivered by Lay Counselor | Enhanced Usual Care
Number analyzed (Participants) | 25 | 25 | 24
score on a scale | -24.2 (25.8) | -23.5 (30.2) | -13.4 (25.4)

10. Secondary Outcome: Mean Depressive Disorder Score Among Participants
Description: Depression symptoms will be evaluated via the 21-item Depression, Anxiety, and Stress Scale (DASS-21), which consists of three subscales. Responses are ranked from 0 (Does not apply to me at all) to 3 (Applied to me very much or most of the time). All subscales are multiplied by 2. Scores on the depression subscale range from 0-42, with ≥ 14 on the depression subscale indicating a depressive disorder.
Time Frame: 6 weeks after enrollment
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Friendship Bench Delivered by Professional Counselor | Friendship Bench Delivered by Lay Counselor | Enhanced Usual Care
Number analyzed (Participants) | 25 | 25 | 24
score on a scale | 8.2 (12.3) | 6.2 (7.4) | 9.0 (9.1)

11. Secondary Outcome: Absolute Reduction in Depressive Symptoms
Description: The absolute reduction of depressive symptoms from baseline to 6 weeks will be evaluated via the DASS-21 depression subscale. Depression symptoms will be evaluated via the 21-item Depression, Anxiety, and Stress Scale (DASS-21), which consists of three subscales. Responses are ranked from 0 (Does not apply to me at all) to 3 (Applied to me very much or most of the time). All subscales are multiplied by 2. Scores on the depression subscale range from 0-42, with ≥ 14 on the depression subscale indicating a depressive disorder.
Time Frame: 6 weeks after enrollment
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Friendship Bench Delivered by Professional Counselor | Friendship Bench Delivered by Lay Counselor | Enhanced Usual Care
Number analyzed (Participants) | 25 | 25 | 24
score on a scale | -8.2 (10.6) | -7.8 (10.5) | -5.4 (10.7)

12. Secondary Outcome: Mean Anxiety Disorder Score Among Participants
Description: Anxiety symptoms will be evaluated via the 21-item Depression, Anxiety, and Stress Scale (DASS-21), which consists of three subscales. Responses are ranked from 0 (Does not apply to me at all) to 3 (Applied to me very much or most of the time). All subscales are multiplied by 2. Scores on the anxiety subscale range from 0-42, with ≥ 10 on the anxiety subscale indicating an anxiety disorder.
Time Frame: 6 weeks after enrollment
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Friendship Bench Delivered by Professional Counselor | Friendship Bench Delivered by Lay Counselor | Enhanced Usual Care
Number analyzed (Participants) | 25 | 25 | 24
score on a scale | 8.2 (8.3) | 8.3 (8.7) | 11.0 (7.9)

13. Secondary Outcome: Absolute Reduction in Anxiety Symptoms
Description: The absolute reduction of anxiety symptoms from baseline to 6 weeks will be evaluated via the DASS-21 anxiety subscale. Anxiety symptoms will be evaluated via the 21-item Depression, Anxiety, and Stress Scale (DASS-21), which consists of three subscales. Responses are ranked from 0 (Does not apply to me at all) to 3 (Applied to me very much or most of the time). All subscales are multiplied by 2. Scores on the anxiety subscale range from 0-42, with ≥ 10 on the anxiety subscale indicating an anxiety disorder.
Time Frame: 6 weeks after enrollment
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Friendship Bench Delivered by Professional Counselor | Friendship Bench Delivered by Lay Counselor | Enhanced Usual Care
Number analyzed (Participants) | 25 | 25 | 24
score on a scale | -6.4 (6.7) | -5.9 (10.6) | -3.9 (9.4)

14. Secondary Outcome: Mean Stress Disorder Score Among Participants
Description: Stress symptoms will be evaluated via the 21-item Depression, Anxiety, and Stress Scale (DASS-21), which consists of three subscales. Responses are ranked from 0 (Does not apply to me at all) to 3 (Applied to me very much or most of the time). All subscales are multiplied by 2. Scores on the stress subscale range from 0-42, with ≥ 19 on the stress subscale indicating a stress disorder.
Time Frame: 6 weeks after enrollment
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Friendship Bench Delivered by Professional Counselor | Friendship Bench Delivered by Lay Counselor | Enhanced Usual Care
Number analyzed (Participants) | 25 | 25 | 24
score on a scale | 10.9 (9.8) | 9.4 (8.2) | 12.3 (7.8)

15. Secondary Outcome: Absolute Reduction in Stress Symptoms
Description: The absolute reduction of stress symptoms from baseline to 6 weeks will be evaluated via the DASS-21 stress scale. Stress symptoms will be evaluated via the 21-item Depression, Anxiety, and Stress Scale (DASS-21), which consists of three subscales. Responses are ranked from 0 (Does not apply to me at all) to 3 (Applied to me very much or most of the time). All subscales are multiplied by 2. Scores on the stress subscale range from 0-42, with ≥ 19 on the stress subscale indicating a stress disorder.
Time Frame: 6 weeks after enrollment
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Friendship Bench Delivered by Professional Counselor | Friendship Bench Delivered by Lay Counselor | Enhanced Usual Care
Number analyzed (Participants) | 25 | 25 | 24
score on a scale | -9.5 (11.1) | -9.8 (11.9) | -4.1 (10.2)

16. Secondary Outcome: Mean Proportion of Days With MMT Adherence
Description: Out of the first 183 days of study participation, the total number of days a participant attended their MMT visit appointment divided by 183 days.
Time Frame: Study baseline through 6 months of follow-up
Population: The analysis population includes the number of participant MMT visits for all participants who had complete MMT adherence data from baseline to 6 months (183 days in total). All participants (n=25) in each intervention arm had complete data for a total of 4575 (25*183) visits, while n=23 participants in the usual care arm had complete data for a total of 4209 (23*183) visits. Note: data was collected at the participant level.
Measure: Mean (Standard Deviation); unit: proportion of days
Units Other Than Participants: MMT visits
Arm/Group | Friendship Bench Delivered by Professional Counselor | Friendship Bench Delivered by Lay Counselor | Enhanced Usual Care
Number analyzed (Participants) | 25 | 25 | 23
Number analyzed (MMT visits) | 4575 | 4575 | 4209
proportion of days | 0.99 (0.03) | 0.99 (0.01) | 0.96 (0.14)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of signing informed consent through completion of the follow up period, a total of 1 year.
Arm/Group | Friendship Bench Delivered by Professional Counselor | Friendship Bench Delivered by Lay Counselor | Enhanced Usual Care
All-Cause Mortality (participants affected / at risk) | 0/26 | 1/25 | 0/26
Serious Adverse Events (participants affected / at risk) | 1/26 | 0/25 | 0/26
Other Adverse Events (participants affected / at risk) | 2/26 | 1/25 | 0/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Friendship Bench Delivered by Professional Counselor (N=26) | Friendship Bench Delivered by Lay Counselor (N=25) | Enhanced Usual Care (N=26)
Pancreatitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Friendship Bench Delivered by Professional Counselor (N=26) | Friendship Bench Delivered by Lay Counselor (N=25) | Enhanced Usual Care (N=26)
Suicidal Thoughts / Ideations (Psychiatric disorders) | 2 (2) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-10-01): https://cdn.clinicaltrials.gov/large-docs/01/NCT04790201/Prot_SAP_001.pdf
  • Informed Consent Form (2022-04-01): https://cdn.clinicaltrials.gov/large-docs/01/NCT04790201/ICF_000.pdf